CLINICAL TRIAL: NCT02018965
Title: Role of Extended-release Niacin on Immune Activation in HIV-infected Patients Treated With Antiretroviral Therapy: a Proof-of-concept Study
Brief Title: Niacin on Immune Activation : a Proof-of-concept Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Dr. Bertrand Lebouche, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTN006
Record Dates: First submitted 2013-12-17; First posted 2013-12-24 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: HIV
Keywords: HIV; Extended-release Niacin; Immune activation
MeSH Terms: interventions — Niacin; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ER niacin followed by ART alone (Other): For Arm 1, ER niacin administration begins Week 0 and ends Week 24 (defined as 'immediate use' arm).
  Interventions: Drug: Niacin
- ART alone followed by ER niacin (Other): For Arm 2, ER niacin administration begins after the Week 24 Visit and ends Week 48 (defined as 'deferred use' arm).
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Niacin — • Group 1: This group will receive an initial dose of ER niacin 500 mg by mouth, the first evening from week 0 to week 4 then increase it to 1000 mg once a day from week 5 to week 8, then increase to 1500 mg from week 9 to week 12 then increase to 2000 mg until weeks 24 and then stopped.
  Participants will continue to take their ART treatment as prescribed throughout the study.
  Other Names: Niaspan FCT®; extended-release(ER)Niacin; vitamin B3
Drug: Niacin — • Group 2: This group will not receive ER niacin for the first 24 weeks. This group will receive an initial dose of ER niacin 500 mg the first evening at week 25 by mouth from week 25 to week 28 then increase it to 1000 mg once a day from week 29 to week 32, then increase to 1500 mg from week 33 to week 36 then increase to 2000 mg until week 48 and then stopped.
  Participants will continue to take their ART treatment as prescribed throughout the study.
  Other Names: Niaspan FCT®; extended-release(ER)Niacin; vitamin B3

SUMMARY:
There are a number of powerful anti-HIV drugs, which keep the virus at undetectable levels and enable HIV-infected individuals to live longer. However, some participants taking anti-HIV drugs do not achieve an adequate CD4 recovery and remain at risk for developing AIDS and non-AIDS-related complications.

ER niacin (PrNiaspanFCT®) is an extended-released form of niacin, also known as vitamin B3. Niacin is effective in reducing cholesterol levels in the blood. This drug has been known for a long-time to treat dyslipidemia and it is used to improve favourably all the lipoprotein risk factors for artherosclerotic disease, particularly in HIV-infected patients. Recent scientific research shows that regular consumption of niacin-rich foods may also provide protection against Alzheimer's disease and age-related cognitive decline.

The purpose of this study is to find out:

1. If ER niacin combined with anti-HIV drugs, compared with anti-HIV drugs alone, could reduce T cell immune activation and enhance CD4 recovery;
2. If ER niacin can improve your quality of life and your neurocognitive functions

DETAILED DESCRIPTION:
Primary objective

• To assess the impact of extended-release niacin (ER niacin) supplementation + antiretroviral therapy (ART) compared to ART alone on T-cell immune activation as defined by CD8CD38 percentage

Secondary objectives

* To assess the change in total CD4 T-cell count after ER niacin administration
* To explore the effect of ER niacin on regulatory T-cells (Th-17/Treg) in blood and gut mucosa samples
* To explore the effect of ER niacin on cytokines and inflammatory markers such as INF-α, IL-1, IL-6, IL-17, D-dimers, usCRP and LPS
* To assess the influence of ER niacin on tryptophan (Trp) plasmatic levels
* To assess changes in cholesterol and triglycerides
* To explore ER niacin tolerance
* To evaluate the impact of ER niacin on quality of life (QoL), fatigue, depression, and neurocognitive scores

Population: All participants will have an undetectable HIV viral load (< 50 copies/mL) for at least 3 months, current CD4 cell count of < 350 cells/µL and be receiving ART for at least the previous 12 months.

Sample size: N=20

ELIGIBILITY:
Participants must meet all of the following criteria within four weeks prior to the Week 0 (Baseline) Visit to be considered eligible for entry into the study:

1. Documented HIV infection by Western Blot, EIA assays or viral load assay
2. Aged 21 or older
3. Viral load < 50 copies/mL for the last 3 months
4. CD4 cell count < 350 cells/µL
5. On stable ART, i.e., ART unchanged for treatment failure (rebound in viral load) for more than 12 months
6. Able to communicate adequately in either French or English
7. Able and willing to give written informed consent prior to enrolment including access to relevant medical records.

Participants are not eligible to participate in the study if any of the following conditions are met:

1. Pregnant, breastfeeding or planning to become pregnant during the course of the study. All fecund female participants must undergo a pregnancy test, with a negative result, prior to being eligible to participate in the study
2. Prior history of hypersensitivity reaction to niacin or any other component of the study drug
3. Prior history of flushing
4. Active liver disease or unexplained persistent elevations of serum transaminases
5. Co-infection with active Hepatitis B or C virus (positive HBs Ag or positive anti HBc antibodies with a detectable HBV DNA viral load or positive anti HCV antibodies with a detectable HCV RNA viral load)
6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or alkaline phosphatase >2.5 x upper limit of normal (ULN)
7. Active duodenal or gastric peptic ulcer
8. Active bleeding disorders
9. History of gout
10. Active AIDS events in the last 3 months as determined by the treating physician
11. Unstable angina or acute phase myocardial infarction, with or without vasodilator agents
12. Diabetic or potentially diabetic with hypercholesterolaemia
13. Renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in CD8CD38 percentage | 24 weeks
  Comparison of the change in CD8CD38 percentage from Week 0 to Week 24 of Arm 1 (ER niacin + ART) to Week 0 to Week 24 of Arm 2 (ART alone) (ER niacin treatment + ART vs. ART alone for 24 weeks)
Comparison of the change in CD8CD38 percentage during the ER niacin + ART period | 48 weeks
  Comparison of the change in CD8CD38 percentage during the ER niacin + ART period with the change in CD8CD38 during the ART alone period within each arm (Week 0 to Week 24 vs. Week 24 to Week 48 for Arm 1 and Week 24 to Week 48 vs. Week 0 to Week 24 for Arm 2); if the difference between ER niacin versus control is similar in the two time periods, the treatment effect will be pooled adjusting for treatment order

SECONDARY OUTCOMES:
Change in CD4 cell count and their subsets, including naïve, central memory and effector memory and Th17/Treg cells | 48 weeks
Changes in inflammatory markers such as INF-α, IL-1, IL-6, IL-17, usCRP, LPS and D-dimers | 48 weeks
Change in plasmatic Trp levels | 48 weeks
Changes in total cholesterol, HDL, LDL cholesterol and triglycerides | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lebouche B, Jenabian MA, Singer J, Graziani GM, Engler K, Trottier B, Thomas R, Brouillette MJ, Routy JP. The role of extended-release niacin on immune activation and neurocognition in HIV-infected patients treated with antiretroviral therapy - CTN PT006: study protocol for a randomized controlled trial. Trials. 2014 Oct 7;15:390. doi: 10.1186/1745-6215-15-390. PMID 25293882